CLINICAL TRIAL: NCT04855552
Title: Pilot Telehealth Weight Loss Program for Breast Cancer Survivors
Brief Title: Telehealth Weight Loss Program for Breast Cancer Survivors
Acronym: TWL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Julia Tchou, Co-Director of the Rena Rowan Breast Center, Director of Breast Cancer Immuno-Oncology Research, Professor of Clinical Surgery, and Principal Investigator, Abramson Cancer Center at Penn Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 17120; 844762 (Other: IRB)
Record Dates: First submitted 2021-04-08; First posted 2021-04-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cancer Survivors; Cancer of Breast; Body Weight; Overweight and Obesity
Keywords: Breast Cancer; Cancer Survivor; Body Mass Index; Telehealth; Breast Carcinoma; Overweight; Obese
MeSH Terms: conditions — Breast Neoplasms; Body Weight; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Single-arm longitudinal group to examine patient-reported outcomes, body mass, and mammographic density changes pre-and post-intervention.
Masking Description: 12 patients (and possibly up to 20) (2 telehealth groups with at least 6 participants; 1 group leader per group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arms Longitudinal Group (Experimental): Behavioral weight-loss program via telehealth (video conferencing). Participants will receive weekly group sessions of lifestyle counseling for the first 20-weeks, followed by every other week sessions in weeks 22 and 24, for a total of 6-months of intervention.
  Interventions: Behavioral: Behavioral Weight-loss Program Via Telehealth; Behavioral: Behavioral Weight-Loss Program Via Telehealth - Weight Measures; Behavioral: Validated Surveys of Patient-Reported Outcomes

INTERVENTIONS:
Behavioral: Behavioral Weight-loss Program Via Telehealth — Investigators will use a manual based on the DPP, as adapted previously for the endometrial cancer population and now adapted for breast cancer survivors. Dr.Courtney McCuen-Wurst, has extensive experience in working with persons with overweight and obesity with medical comorbidities. She also has experience leading group interventions at our Center via telehealth. The content of the sessions addresses the domains associated with behavioral weight management including nutrition, exercise, stress and emotion management, and lifestyle modification strategies (to improve adherence to the diet and activity plan). Participants will monitor energy intake and physical activity daily to help them achieve recommended calorie and activity goals. Self-monitoring will be encouraged online with MyFitnessPal.com, which will be shared with the study staff to increase accountability and provide opportunity for feedback to participants.
Behavioral: Behavioral Weight-Loss Program Via Telehealth - Weight Measures — Each participant will also be mailed a digital scale (Eat Smart) so they can weigh themselves each week and report their weight to the group leader; patients will be encouraged to take a picture of their weight on the scale after they step off (the number remains for 3-seconds) and send the picture to Dr. McCuen-Wurst. Participants will be encouraged to start with at least 1-minutes of moderately vigorous physical activity (e.g. brisk walking, swimming), at least five days per week, building up to at least 30-minutes per day (150-minutes per week) by week-6.
Behavioral: Validated Surveys of Patient-Reported Outcomes — The following surveys will be completed by participants pre- and post-intervention:
  * COH-QOL Instrument - Breast Cancer Patient (QOL-BC)
  * International Physical Activity Questionnaire (IPAQ) Short Form
  * Patient Health Questionnaire (PHQ-9) (Depression)
  * Acceptability of Intervention Measure
  The following survey will be completed post-intervention
  • Exit interview regarding acceptability of the program.
  The following measurements/clinical tests results will be collected and compared pre- and post-intervention:
  * Anthropometric measurements: height (self-report); weight (as measured on scale provided by study)
  * Mammographic breast density estimated in annual clinical mammogram

SUMMARY:
This is a single-arm longitudinal group to examine patient-reported outcomes, body mass and mammographic density changes pre- and post- weight loss intervention of breast cancer survivors using video conferencing telehealth visits.

DETAILED DESCRIPTION:
Participants will receive weekly group sessions of lifestyle counseling for the first 20 weeks, followed by every other week sessions in weeks 22 and 24, for a total of 6 months of intervention. These group sessions, with 6 participants per group, will be delivered virtually via a HIPAA Compliant Teleconference Platform. The expected number of participants is at least 2 and no more than 6 in this 90-min group sessions which will be provided by a counselor from Penn Center for Weight and Eating Disorders.

The content of the sessions addresses the domains associated with behavioral weight management, including nutrition, exercise, stress and emotion management, and lifestyle modification strategies (to improve adherence to the diet and activity plan). Participants will monitor energy intake and physical activity daily to help them achieve recommended calorie and activity goals. Self-monitoring will be encouraged online with MyFitnessPal.com, which will be shared with the study staff to increase accountability and provide opportunity for feedback to participants.

Each participant will also be mailed a digital scale so they can weigh themselves each week and report their weight to the group leader. Participants will be encouraged to start with at least 10 minutes of moderately vigorous physical activity (e.g., brisk walking, swimming), at least five days per week, building up to at least 30 minutes per day (150 minutes per week) by week 6.

The primary objective is to assess feasibility and acceptance of telehealth weight loss intervention by the participants. The participants will be asked to complete the following surveys at two time points: baseline (pre-) and treatment end (at week 24). The participants will complete the following psychosocial measures.

1. City of Hope Quality of Life (COH-QOL) Instrument - Breast Cancer Patient (QOL-BC)
2. The International Physical Activity Questionnaire (IPAQ) Short Form - that assess the types and intensity of physical activity and sitting time in which people routinely engage. It provides an estimate of total physical activity in MET-min/week and time spent sitting.
3. Patient Health Questionnaire (PHQ-9) (Depression)
4. Acceptability of Intervention Measure

Finally, investigators will conduct an exit interview with each participant to assess the acceptability of the intervention, the delivery of the intervention via telehealth, and the patients' satisfaction with their treatment outcomes. Investigators will also solicit suggestions for improvements to the program for future interventions.

The secondary objectives are to measure changes from pre- to post weight-loss intervention for 1) body mass and 2) mammographic breast density.

To assess body mass changes, weight will be reported at baseline and after week 24 of the intervention. The scale will be mailed to participants at the beginning of the study. Participants' height from the electronic medical record will be used. Percent weight loss will be calculated to assess weight change across participants.

To assess mammographic breast density changes, investigators will measure mammographic density of annual mammogram pre- and post weight-loss program. Annual mammograms are routinely performed for breast cancer survivors except for those who have had bilateral mastectomy. Two annual mammograms will be used to measure mammographic density. The annual mammogram performed between 1 month - 12 months prior to weight loss program initiation will be used as baseline (pre-intervention). The post-intervention mammogram will be the first annual mammogram performed after weight loss program. If routine annual mammogram occurs during the 20-week weight loss program, then the next annual mammogram will be used for breast density assessment.

Therefore, study duration for each participant from enrollment to completion (mammographic density) is estimated to be up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* History of in situ or invasive breast cancer
* Have completed breast cancer surgery, adjuvant cytotoxic chemotherapy (as indicated) and adjuvant radiation therapy (as indicated) at least 6-months prior to enrollment
* Not on active treatment for other cancer for at least 6-months prior to enrollment
* Currently cancer free
* Overweight or obese (BMI of 25 kg/m^2 or greater)
* Have internet access and videoconferencing capability

Exclusion Criteria:

* Current use of weight loss medication (OTC or prescription) or participation in behavioral weight loss program
* Currently participating in a behavioral weight loss program
* Self-report of alcohol or substance abuse within the past 12-months, including at-risk drinking (current consumption of more than 14 drinks per week)
* Undergone bilateral mastectomy
* History of Bulimia nervosa
* Inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine feasibility and Acceptability Using the City of Hope Quality of Life Instrument - Breast Cancer Patient to Assess Changes in Quality of Life | 24 weeks
  To determine the feasibility and acceptability of a weight loss program via telehealth for breast cancer survivors. The participants will be asked to complete the City of Hope Quality of Life Instrument (COH-QOL) - Breast Cancer Patient (QOL-BC) at two time points: baseline (pre-) and treatment end (at week 24).
  * COH-QOL Instrument - Breast Cancer Patient (QOL-BC) - 46 items
  * The scoring is based on a scale of 0 = worst outcome to 10 = best outcome. Some items have reverse anchors and the value should be scored as the reverse of the item circled, e.g., if a patient selected "4" then their score on a reverse anchor would be 10 - 4 = 6.
Determine feasibility and Acceptability Using the International Physical Activity Questionnaire to Assess Changes in Physical Activity | 24 weeks
  To determine the feasibility and acceptability of a weight loss program via telehealth for breast cancer survivors. The participants will be asked to complete the International Physical Activity Questionnaire (IPAQ) at two time points: baseline (pre-) and treatment end (at week 24).
  * The International Physical Activity Questionnaire (IPAQ) Short Form
  * This is an open-ended questionnaire surrounding individuals' last 7-day recall of physical activity.
Determine feasibility and Acceptability Using the Patient Health Questionnaire to Assess Changes in Measures of Depression | 24 weeks
  To determine the feasibility and acceptability of a weight loss program via telehealth for breast cancer survivors. The participants will be asked to complete the Patient Health Questionnaire (PHQ-9) (Depression) at two time points: baseline (pre-) and treatment end (at week 24).
  - The PHQ-9 is a nine item questionnaire and the scoring is based on a scale of 0= best outcome to 3 = worst outcome. Total scores range from 0 to 27 and higher scores are associated with higher severities of depression, ranging from minimal to severe.
Using the Acceptability of Intervention Measure to Assess Acceptability and Feasibility | 24 weeks
  To determine the feasibility and acceptability of a weight loss program via telehealth for breast cancer survivors. The participants will be asked to complete the Acceptability of Intervention Measure at two time points: baseline (pre-) and treatment end (at week 24).
  - The Acceptability of Intervention Measure is a four item questionnaire and the scoring is based on a scale ranging from 1 = completely disagree to 5= Completely Agree. Higher scores are associated with greater acceptability of the intervention.
Requesting Direct Verbal Feedback From Participants to Assess Elements of the Program that Work Well, to Acquire Suggestions, and to Seek Suggestions to Determine Feasibility and Acceptability | 24 weeks
  Finally, investigators will conduct an exit interview with each participant to assess the acceptability of the intervention, the delivery of the intervention via telehealth, and their satisfaction with their treatment outcomes. Investigators will also solicit suggestions for improvements to the program for future interventions.

SECONDARY OUTCOMES:
To measure changes from pre- to post-weight-loss intervention for 1) body mass. | 24 Months
  To assess change in body mass index (BMI), height (measured in meters) and weight (measured in kilograms) will be combined to report BMI in kg/m^2. Weight will be reported at baseline and after week 24 of the intervention. Participants' height (in meters) will be collected from the electronic medical record at baseline.
To measure changes from pre- to post-weight-loss intervention for 2) Qualitative Changes in Mammographic Breast Density | 24 Months
  To assess mammographic breast density changes, investigators will measure mammographic density of annual mammogram pre- and post-weight-loss program. The qualitative MBD as reported by Breast Imaging-Reporting and Data System (BI-RADS) scores are collected from the clinical radiologist reports.
To measure changes from pre- to post-weight-loss intervention for 2) Quantitative Changes in Mammographic Breast Density | 24 months
  To assess mammographic breast density changes, investigators will measure mammographic density of annual mammogram pre- and post-weight-loss program. Quantitative MBD will be analyzed using LIBRA, which is a fully-automated, free, and publicly available program that estimates MBD. Following digital segmentation, the LIBRA software analysis provides breast area, absolute dense area, and area percent density for each image of a mammographic study. Mean breast area (cm^2), mean dense area (cm^2), and quantitative MBD (%) will be calculated for each mammographic study as described.

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Tchou, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania (Hospital of the University of Pennsylvania), Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Goodwin PJ, Segal RJ, Vallis M, Ligibel JA, Pond GR, Robidoux A, Findlay B, Gralow JR, Mukherjee SD, Levine M, Pritchard KI. The LISA randomized trial of a weight loss intervention in postmenopausal breast cancer. NPJ Breast Cancer. 2020 Feb 21;6:6. doi: 10.1038/s41523-020-0149-z. eCollection 2020. PMID 32133391
- [Background] Ligibel JA, Barry WT, Alfano C, Hershman DL, Irwin M, Neuhouser M, Thomson CA, Delahanty L, Frank E, Spears P, Paskett ED, Hopkins J, Bernstein V, Stearns V, White J, Hahn O, Hudis C, Winer EP, Wadden TA, Goodwin PJ. Randomized phase III trial evaluating the role of weight loss in adjuvant treatment of overweight and obese women with early breast cancer (Alliance A011401): study design. NPJ Breast Cancer. 2017 Sep 21;3:37. doi: 10.1038/s41523-017-0040-8. eCollection 2017. PMID 28948213
- [Background] Krouse RS, Grant M, McCorkle R, Wendel CS, Cobb MD, Tallman NJ, Ercolano E, Sun V, Hibbard JH, Hornbrook MC. A chronic care ostomy self-management program for cancer survivors. Psychooncology. 2016 May;25(5):574-81. doi: 10.1002/pon.4078. Epub 2016 Jan 25. PMID 26804708
- [Background] Williams AD, So A, Synnestvedt M, Tewksbury CM, Kontos D, Hsiehm MK, Pantalone L, Conant EF, Schnall M, Dumon K, Williams N, Tchou J. Mammographic breast density decreases after bariatric surgery. Breast Cancer Res Treat. 2017 Oct;165(3):565-572. doi: 10.1007/s10549-017-4361-y. Epub 2017 Jun 28. PMID 28660430
- [Background] Eliassen AH, Colditz GA, Rosner B, Willett WC, Hankinson SE. Adult weight change and risk of postmenopausal breast cancer. JAMA. 2006 Jul 12;296(2):193-201. doi: 10.1001/jama.296.2.193. PMID 16835425
- [Background] Parker ED, Folsom AR. Intentional weight loss and incidence of obesity-related cancers: the Iowa Women's Health Study. Int J Obes Relat Metab Disord. 2003 Dec;27(12):1447-52. doi: 10.1038/sj.ijo.0802437. PMID 14634673
- [Background] Birks S, Peeters A, Backholer K, O'Brien P, Brown W. A systematic review of the impact of weight loss on cancer incidence and mortality. Obes Rev. 2012 Oct;13(10):868-91. doi: 10.1111/j.1467-789X.2012.01010.x. Epub 2012 Jun 4. PMID 22672203
- [Background] Howell A, Anderson AS, Clarke RB, Duffy SW, Evans DG, Garcia-Closas M, Gescher AJ, Key TJ, Saxton JM, Harvie MN. Risk determination and prevention of breast cancer. Breast Cancer Res. 2014 Sep 28;16(5):446. doi: 10.1186/s13058-014-0446-2. PMID 25467785
- [Background] Hardefeldt PJ, Penninkilampi R, Edirimanne S, Eslick GD. Physical Activity and Weight Loss Reduce the Risk of Breast Cancer: A Meta-analysis of 139 Prospective and Retrospective Studies. Clin Breast Cancer. 2018 Aug;18(4):e601-e612. doi: 10.1016/j.clbc.2017.10.010. Epub 2017 Oct 17. PMID 29223719
- [Background] van den Brandt PA, Schulpen M. Mediterranean diet adherence and risk of postmenopausal breast cancer: results of a cohort study and meta-analysis. Int J Cancer. 2017 May 15;140(10):2220-2231. doi: 10.1002/ijc.30654. Epub 2017 Mar 5. PMID 28260236
- [Background] Christou NV, Lieberman M, Sampalis F, Sampalis JS. Bariatric surgery reduces cancer risk in morbidly obese patients. Surg Obes Relat Dis. 2008 Nov-Dec;4(6):691-5. doi: 10.1016/j.soard.2008.08.025. Epub 2008 Sep 20. PMID 19026373
- [Background] Adams TD, Stroup AM, Gress RE, Adams KF, Calle EE, Smith SC, Halverson RC, Simper SC, Hopkins PN, Hunt SC. Cancer incidence and mortality after gastric bypass surgery. Obesity (Silver Spring). 2009 Apr;17(4):796-802. doi: 10.1038/oby.2008.610. Epub 2009 Jan 15. PMID 19148123
- [Background] Sjostrom L, Gummesson A, Sjostrom CD, Narbro K, Peltonen M, Wedel H, Bengtsson C, Bouchard C, Carlsson B, Dahlgren S, Jacobson P, Karason K, Karlsson J, Larsson B, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on cancer incidence in obese patients in Sweden (Swedish Obese Subjects Study): a prospective, controlled intervention trial. Lancet Oncol. 2009 Jul;10(7):653-62. doi: 10.1016/S1470-2045(09)70159-7. Epub 2009 Jun 24. PMID 19556163
- [Background] Ursin G, Quershi SA. Mammographic density - a useful biomarker for breast cancer risk in epidemiologic studies. Norsk Epidemiologi. 2009, 10: 59-68.
- [Background] Casagrande DS, Rosa DD, Umpierre D, Sarmento RA, Rodrigues CG, Schaan BD. Incidence of cancer following bariatric surgery: systematic review and meta-analysis. Obes Surg. 2014 Sep;24(9):1499-509. doi: 10.1007/s11695-014-1276-0. PMID 24817500
- [Background] Wijesooriya NR, Mishra V, Brand PLP, Rubin BK. COVID-19 and telehealth, education, and research adaptations. Paediatr Respir Rev. 2020 Sep;35:38-42. doi: 10.1016/j.prrv.2020.06.009. Epub 2020 Jun 18. PMID 32653468
- [Background] Wosik J, Fudim M, Cameron B, Gellad ZF, Cho A, Phinney D, Curtis S, Roman M, Poon EG, Ferranti J, Katz JN, Tcheng J. Telehealth transformation: COVID-19 and the rise of virtual care. J Am Med Inform Assoc. 2020 Jun 1;27(6):957-962. doi: 10.1093/jamia/ocaa067. PMID 32311034
- [Background] Sun V, Ercolano E, McCorkle R, Grant M, Wendel CS, Tallman NJ, Passero F, Raza S, Cidav Z, Holcomb M, Weinstein RS, Hornbrook MC, Krouse RS. Ostomy telehealth for cancer survivors: Design of the Ostomy Self-management Training (OSMT) randomized trial. Contemp Clin Trials. 2018 Jan;64:167-172. doi: 10.1016/j.cct.2017.10.008. Epub 2017 Oct 16. PMID 29051047
- [Background] The Diabetes Prevention Program Research Group. The Diabetes Prevention Program: baseline characteristics of the randomized cohort. The Diabetes Prevention Program Research Group. Diabetes Care. 2000 Nov;23(11):1619-29. doi: 10.2337/diacare.23.11.1619. PMID 11092283
- [Background] Haggerty AF, Hagemann A, Barnett M, Thornquist M, Neuhouser ML, Horowitz N, Colditz GA, Sarwer DB, Ko EM, Allison KC. A Randomized, Controlled, Multicenter Study of Technology-Based Weight Loss Interventions among Endometrial Cancer Survivors. Obesity (Silver Spring). 2017 Nov;25 Suppl 2(Suppl 2):S102-S108. doi: 10.1002/oby.22021. PMID 29086522
- [Background] Keller BM, Chen J, Daye D, Conant EF, Kontos D. Preliminary evaluation of the publicly available Laboratory for Breast Radiodensity Assessment (LIBRA) software tool: comparison of fully automated area and volumetric density measures in a case-control study with digital mammography. Breast Cancer Res. 2015 Aug 25;17:117. doi: 10.1186/s13058-015-0626-8. PMID 26303303
- [Background] Keller BM, Nathan DL, Wang Y, Zheng Y, Gee JC, Conant EF, Kontos D. Estimation of breast percent density in raw and processed full field digital mammography images via adaptive fuzzy c-means clustering and support vector machine segmentation. Med Phys. 2012 Aug;39(8):4903-17. doi: 10.1118/1.4736530. PMID 22894417
- [Background] Analytics, C.f.B.I.C.a. The Laboratory for Individualized Breast Radiodensity Assessment. 2014.
- [Derived] Allison KC, McCuen-Wurst C, Raevsky A, Holmes N, Goldbach M, Guerra CE, Rendle KA, Cadet TJ, Krouse RS, Tchou J. The Group-basEd Telehealth behavioral WEight Loss Program Among Breast Cancer Survivors: A Pilot and Feasibility Study. Obes Sci Pract. 2024 Dec 21;10(6):e70023. doi: 10.1002/osp4.70023. eCollection 2024 Dec. PMID 39713088
- [Derived] Burkbauer L, Goldbach M, Huang C, Lewandowski J, Krouse R, Allison K, Tchou J. Awareness of link between obesity and breast cancer risk is associated with willingness to participate in weight loss intervention. Breast Cancer Res Treat. 2022 Aug;194(3):541-550. doi: 10.1007/s10549-022-06546-y. Epub 2022 Jun 25. PMID 35751715